CLINICAL TRIAL: NCT05194826
Title: Vestibular Socket Therapy Using Fascia Lata Membrane Versus Connective Tissue Graft in Immediate Implants of Aesthetic Zone
Brief Title: Using Fascia Lata Membrane Versus Connective Tissue Graft in Immediate Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VST_21_22
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Connective Tissue Graft; Anterior Aesthetic Zone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia lata membrane (Experimental)
  Interventions: Procedure: Test
- Connective tissue graft both with xenogenic lamina membrane (Active Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Test — immediate implant and VST with fascia lata membrane + xenogenic lamina membrane and particulate bone graft composed of autogenous cortical chips harvested from the surgical site
  Arms: Fascia lata membrane
Procedure: Control — immediate implant and VST with connective tissue graft + xenogenic lamina membrane and particulate bone graft composed of autogenous cortical chips harvested from the surgical site
  Arms: Connective tissue graft both with xenogenic lamina membrane

SUMMARY:
The aim of this study is to evaluate and compare the Vestibular Socket Therapy (VST) technique using fascia lata membrane versus connective tissue graft both with xenogenic lamina membrane in immediate implants of anterior aesthetic zone.

ELIGIBILITY:
Inclusion Criteria:

* Class II socket according to Elian et al, described as facial soft tissue is present but the buccal plate is partially missing following extraction of the tooth in the maxillary anterior region.
* Thin gingival phenotype.
* Bone quality ranges from D2-D3 as gained from preoperative cone-beam computed tomography.
* Presence of at least 3 mm of keratinized gingiva.
* Optimal compliance as evidenced by no missing treatment appointments and a positive attitude towards oral hygiene

Exclusion Criteria:

* Medically compromised patients and systemic conditions precluding implant and periodontal surgery.
* Smokers, diabetics, pregnant or lactating women.
* History of chemotherapy, radiotherapy in head and/or neck region.
* Bisphosphonate therapy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in peri-implant mucosal level | at baseline, 6 months and 12 months
  The changes in peri-implant mucosal level will be assessed by superimposition of scanning files of different intervals to monitor the changes in surface area calculated by software.
Changes in gingival phenotype | at baseline, 6 months and 12 months
  The changes in gingival phenotype could be assessed at 6 months and 12 months intervals by superimposition of DICOM files on CBCT software.
Chaneg in height of labial (facial) plate of bone | at baseline, 6 months and 12 months
  Cone beam computed tomography (CBCT)
Chaneg in thickness of labial (facial) plate of bone | at baseline, 6 months and 12 months
  Cone beam computed tomography (CBCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt